CLINICAL TRIAL: NCT05273580
Title: Wearable and Patient-reported Outcome-based Continuous Assessment and Support Alerts in Advanced Cancer Patients and Their Carers
Brief Title: Wearable and Patient-reported Outcome-based Continuous Assessment and Support Alerts in Palliative Care
Acronym: wePRO-CASA
Status: Completed | Type: Observational
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Thilo Schuler, Principal Investigator, Royal North Shore Hospital
Other Study IDs: wePRO-CASA
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Palliative Care; Wearable Electronic Devices; Patient Reported Outcome Measures; Cancer; Caregiver; Digital Health
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Eligible patients will be identified by the Nurse Practitioner Cancer & Palliative Care.
  Interventions: Device: Garmin VivoSmart 4; Device: mema - ilumivu
- Carers: The respective carers who are identified by the Nurse Practitioner Cancer & Palliative Care as eligible participants.
  Interventions: Device: Garmin VivoSmart 4; Device: mema - ilumivu

INTERVENTIONS:
Device: Garmin VivoSmart 4 — Wearable sensor to record; sleep, stress, heart rate etc.
Device: mema - ilumivu — mEMA is the a self-service platform running on both iOS and Android that is specifically designed for the administration of mobile Ecological Momentary Assessment or Experience Sampling research studies.

SUMMARY:
Non-professional carers (typically family members) play a critical role in providing adequate home care. This research explores the use of wearable sensors (WS) and electronic patient-reported outcome (ePRO) surveys to monitor stress levels of advanced cancer patient/carer dyads. During wear times, WS-triggered ecological momentary assessments (EMAs) were conducted via short smartphone-based surveys. This pilot study investigates the feasibility of EMAs in community palliative care.

DETAILED DESCRIPTION:
Non-professional carers (typically family members) play a critical role in providing adequate home care along with professional caregivers. However, the physical and emotional toll of caring for a family member can lead to distress and burn out of the carer. The latter often results in the need for temporary or permanent institutional care of the patient. This research explores the feasibility of wearable sensors (WS) and electronic patient-reported outcome (ePRO) surveys to monitor activity patterns and stress levels of advanced cancer patient/caregiver dyads in order to understand their needs better.

Throughout the study, wearable sensors are used to passively record physiological data from patient/carer dyads. During wear times, WS recordings trigger ecological momentary assessments (EMAs) conducted via surveys. This pilot investigates the feasibility and acceptability of EMAs in community palliative care and the potential for incorporating EMA-based interventions into routine care. Future studies may explore the possibility of ecological momentary interventions (EMIs) to trigger just-in-time targeted interventions.

ELIGIBILITY:
Inclusion Criteria:

* Palliative care patient attending at Northern Sydney Cancer Centre, RNSH
* Patient and carer dyad
* Both patient and carer consent
* Patient Karnofsky Performance Scale ≥ 50
* Patient and carer have compatible smart phone

Exclusion Criteria:

• Unwilling or unable to give informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Palliative care patient and their respective carer attending at Northern Sydney Cancer Centre, RNSH.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Wearable compliance | 5 weeks
  Wearable compliance (compliance defined HR signal detected for >=70% of daytime hours between 7:30am to 7:30 pm)

SECONDARY OUTCOMES:
Quantitative and qualitative exploration of EMA/EMI acceptability | 2 hours
  Exploration of EMA/EMI acceptability by patient/carer dyads quantitatively using experience surveys and qualitatively using an (optional) focus group.
Correlative analysis of WS signals and ePRO's | 5 weeks
  Correlative analysis of WS signals and ePRO answers with focus on:
  * Intra-dyadic longitudinal trends (Is there correlation between metrics of a patient and their carer?)
  * EMA trigger incidences and distribution of ePRO-stated trigger reasons including "false alarms" of the whole cohort

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Schuler, Principal Investigator — Royal North Shore Hospital
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided
The results of this trial will be published in a peer reviewed journal. We are targeting high-impact palliative care journals such as 'Palliative Medicine' for publication.

REFERENCES:
- See also: Project website — https://thiloschuler.me/project/casa/